CLINICAL TRIAL: NCT04615468
Title: A Single-arm, Open-label, Multi-center, Phase II Study of TQ-B3525 in Subjects With Relapsed/Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: A Study of TQ-B3525 in Subjects With Relapsed/Refractory Peripheral T-cell Lymphoma（PTCL）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-II-04
Record Dates: First submitted 2020-10-30; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-07

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablets (Experimental): TQ-B3525 tablet administered orally.
  Interventions: Drug: TQ-B3525

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQ-B3525 in subjects with relapse/refactory peripheral T-cell lymphoma who have received at least 1 lines of therapeutic schedules. TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and signed an informed consent form; 2. 18 years and older, Eastern Cooperative Oncology Group(ECOG) performance status score of 0 to 2, life expectancy ≥ 3 months; 3. Diagnosis of peripheral T-cell lymphoma (PTCL); 4. Has received at least one line systemic treatment and disease progression after the last treatment; 5. Has at least one measurable lesion; 6. Adequate organ system function; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

* 1. Other types of T-cell lymphoma; 2. Has central nervous system violation; 3. Has received other PI3K inhibitors or CAR-T treatments; 4. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration; 5. Has type I diabetes or uncontrolled type II diabetes; 6. Has history of interstitial lung disease; 7. Has history of interstitial lung disease; 8. Has multiple factors affecting oral medication; 9. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1; 10. Has received systemic steroid treatment within 7 days before the first dose; 11. Has received other systemic anti-tumor medications within 4 weeks before the first administration, or still within the 5 half-life of the medication, which occurs first; 12. Has active infections which need drug treatment; 13. Has received surgery, or unhealed wounds within 4 weeks before the first administration; 14. Has a history of autologous hematopoietic stem cell transplant within 3 months; 15. Has a history of allogeneic hematopoietic stem cell transplant; 16. Grade II or higher cardiovascular disease within 6 months before the first administration; 17. QTCF > 480ms, left ventricular ejection fraction (LVEF)<50%; 18. Urinary protein ≥ 2 +, and 24-hour urinary protein quantity>1g within 7 days; 19. Has active hepatitis B or C; 20. Has psychotropic substances abuse or a mental disorder; 21.Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) by Independent Review Committee | up to 6 months
  Percentage of participants achieving complete response (CR) and partial response (PR) based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by Investigator | up to 6 months
  Percentage of participants achieving complete response (CR) and partial response (PR) assessed by investigator.
Duration of response (DOR) | up to 12 months
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 6 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Disease control rate（DCR） | up to 12 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall survival(OS) | up to 24 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality